CLINICAL TRIAL: NCT06434779
Title: Single Arm, Multicenter, Prospective Registry Investigating Efficacy and Safety of Mechanical Thrombectomy (JETi®) in Acute and Acute-on-Chronic Arterial Occlusions in Femoro-popliteal and Proximal BTK-Lesions (JETART)
Brief Title: Investigating Efficacy and Safety of JETi® in Arterial Occlusions in FEM-POP and Prox BTK-Lesions (JETART)
Acronym: JETART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Science LP GmbH (Other)
Collaborators: ID3 Medical (Other); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iD320240306
Record Dates: First submitted 2024-03-06; First posted 2024-05-30 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanical Thrombectomy (JETi®) (Experimental)
  Interventions: Device: JETi 6F and 8F Thrombectomy system

INTERVENTIONS:
Device: JETi 6F and 8F Thrombectomy system — To demonstrate the efficacy and safety of the mechanical thrombectomy device (JETi 6F and 8F) for treatment of patients with symptomatic peripheral artery disease (PAD) due to acute or acute on chronic occlusions of the femoral and/or popliteal arteries and the first 10 cm of the below-the -knee arteries.

SUMMARY:
To demonstrate the efficacy and safety of the mechanical thrombectomy device (JETi 6F and 8F) for treatment of patients with symptomatic peripheral artery disease (PAD) due to acute or acute on chronic occlusions of the femoral and/or popliteal arteries and the first 10 cm of the below-the -knee arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years
* Patient has Rutherford Classification 2,3 or 4.
* Patient has provided written informed consent and is willing to comply with study follow-up requirements.

Angiographic inclusion criteria

* De novo thrombotic occlusive lesion(s) or thrombotic re-occlusion or in-stent thrombotic occlusive lesion(s) or thrombotic occlusion of a bypass (autolog or prosthetic) occurring acute or subacute with onset of complains within <30 days prior to first seen by investigating physician.
* Target lesion is located between the ostium of the SFA and the end of the P3 segment of the popliteal artery, tibioperoneal trunk, respectively the first 10 cm of the below the knee vessels
* Target vessel diameter ≥ 3 mm and ≤ 8 mm and irrespective of lesion length
* Target lesion must be occlusive lesion Note: there is no limitation in lesion length
* Successful, uncomplicated crossing of the target lesion occurs when the tip of the guidewire is distal to the target lesion without the occurrence of flow-limiting dissection of perforation and is judged by visual inspection to be within the true lumen.
* A patent inflow artery free from significant stenosis (≥50% stenosis) as confirmed by angiography.
* At least one patent native distal outflow artery to the ankle or foot, free from significant stenosis (≥ 50 % stenosis) as confirmed by angiography.

Exclusion Criteria:

* Patients meets any contraindication for JETi mechanical thrombectomy use per IFU
* Lesion crossing is difficult and the lesion is not suspicious for fresh thrombus containment
* Pregnant women or female patients of childbearing potential that do not use adequate contraceptive methods
* Patient has a life expectancy of less than 1 year
* Patient has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Patient is allergic to all anti-platelet treatments
* Patient has platelet count <100.000/mm3 or >700.000/mm
* Patient has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the study procedure
* Patient is diagnosed with coagulopathy that bares the risk of increased bleeding risk
* Patient has history of stroke within past 90 days
* Patient is participating in an investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study.
* Patient has had any major (e.g. cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure
* Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol
* Patient suffering from HIT II

Angiographic Exclusion Criteria:

* Target lesion is larger than 8 mm, respectively smaller than 3 mm
* Significant target vessel tortuosity or other parameters prohibiting access to the target lesion
* Absence of thrombus in the target vessel
* Iliac inflow disease requiring treatment, unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤ 30 % residual diameter stenosis without death or major complications.
* No patent outflow vessels on the level of 10 cm below the origin of below the-knee arteries to the level of the foot or ankle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | During index procedure
  The primary efficacy endpoint is technical procedural success (post Jeti) defined as restoration of impaired flow to a straight-line orthograde flow in the target vessel/bypass with near complete or complete recanalization of occluded vessel by using the JETI system prior to further additional endovascular therapy.
Primary Safety Endpoint | Up to 30 days post-index procedure
  The primary safety endpoint is a composite of
  1. freedom from device- and procedure-related death through 30 days post-index procedure;
  2. freedom from major target limb amputation (above-the-ankle (ATA)) through 30 days post-procedure and
  3. freedom from clinically-driven target vessel revascularization (CD-TVR) through 30 days post-index procedure

SECONDARY OUTCOMES:
Acute device success | During index procedure
  Defined as successful delivery of the device to the lesion
Secondary safety endpoint at discharge up to 30 days post index procedure | Up to 30 days
  Secondary safety endpoint is a composite of
  1. freedom from Major Adverse Events (MAEs). MAEs are defined as: all-cause death; bleeding, hematoma and intracranial hemorrhage; major target limb amputation; thrombosis at the target lesion.
  2. freedom from major target limb amputation and MALE
  3. freedom from CD-TVR
Sustained clinical improvement at discharge and at 30- days post-index procedure | Hospital admission to discharge up to 30 days and at 30 days
  Clinical improvement is defined as a composite of
  1. freedom from major target limb amputation,
  2. freedom from TVR,
  3. freedom from worsening target limb Rutherford class (compared to baseline)
  4. freedom from decrease in target limb ankle brachial index (ABI) ≥0.15 (compared to baseline)
Primary Patency at discharge and at 30 days post-index procedure | Hospital admission to discharge up to 30 days and at 30 days
  The primary patency is defined as a composite of
  1. freedom from clinically-driven target lesion revascularization (CD-TLR)
  2. freedom from binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis) as confirmed by an independent Corelab
Freedom from TLR at discharge and at 30 days post-index procedure | Hospital admission to discharge up to 30 days and at 30 days
  TLR is defined as a reintervention to maintain or restore the patency in the target lesion. TLR is clinically-driven (CD) when the TLR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
Change in target limb Rutherford Classification from baseline to 30 days post-index procedure | Up to 30 days
  Change in target limb Rutherford Classification from baseline to 30 days post-index procedure
Change in target limb resting ABI from baseline to discharge and at 30 days post-index procedure | Up to 30 days
  Change in target limb resting ABI from baseline to discharge and at 30 days post-index procedure
Change of life quality according to the Walking Impairment Questionnaire (WIQ) from baseline to 30 days post-index procedure | Up to 30 days
  Change of life quality according to the Walking Impairment Questionnaire (WIQ) from baseline to 30 days post-index procedure
Change of life quality according to the EQ-5D questionnaire from baseline to 30 days post-index procedure | Up to 30 days
  Change of life quality according to the EQ-5D questionnaire from baseline to 30 days post-index procedure
Duration of hospital stay | Hospital admission to discharge up to 30 days
  Duration of hospital stay

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan